CLINICAL TRIAL: NCT01998594
Title: Use of FlexHD as a Post-Trapeziectomy Spacer in Patients Treated for Thumb Basal Joint Arthritis
Brief Title: Use of FlexHD as Post Trapeziectomy Spacer
Acronym: MTF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Musculoskeletal Transplant Foundation (Other)
Responsible Party: Principal Investigator, David Kulber, MD, Director Plastic Surgery, Center of Excellence, Cedars Sinai; Clinical Professor of Surgery, USC Keck School of Medicine, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00027968
Record Dates: First submitted 2013-11-13; First posted 2013-12-02 (Estimated); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Osteoarthrosis of the Carpometacarpal Joint of the Thumb
Keywords: Thumb arthritis; CMC arthritis; Arthroplasty
MeSH Terms: interventions — Arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arthroplasty without HADM (Active Comparator): Three - five (3 - 5) subjects with Eaton stage III-IV thumb CMC osteoarthritis undergo the basilar joint arthroplasty procedure without using a spacer constructed from human acellular matrix (HADM). Their postoperative DASH scores, grip strength, pinch strength, pain scale scores and quality of life questionnaires are compared to their preoperative scores. These subjects will be compared with a group of twenty-five (25) similar subjects who received the arthroplasty procedure with the use of the HADM spacer.
  Interventions: Procedure: Arthroplasty
- Arthroplasty with HADM (Experimental): Twent-five (25) subjects with Eaton stage III-IV thumb CMC osteoarthritis undergo the basilar joint arthroplasty procedure with an interposition arthroplasty technique using a spacer constructed from human acellular matrix (HADM). Their postoperative DASH scores, grip strength, pinch strength, pain scale scores and quality of life questionnaires are compared to their preoperative scores. These subjects will be compared with a group of three - five (3 - 5) similar subjects who received the arthroplasty procedure without the use of the HADM spacer.
  Interventions: Procedure: Arthroplasty

INTERVENTIONS:
Procedure: Arthroplasty — A longitudinal dorsoradial incision is made from the base of the first metacarpal to the radial styloid for access to the thumb CMC joint. Trapeziectomy is performed piecemeal using sharp and blunt dissection. The base of the first metacarpal is then decorticated with a sagittal saw. A 4x7 cm sheet of thin FlexHD (HADM) is fashioned by a 4-0 monocryl suture imbrication into the size and shape of the subject's trapezium, keeping the dermal side exposed as much as possible. The allograft is secured with multiple interrupted 3-0 Ticron sutures and the bundle is placed into the post-trapeziectomy space. Additional suture fixation is performed between the FlexHD and the volar capsule of the trapezium, and base of the thumb metacarpal using 4-0 Mersilene sutures. The control treatment group will have the same trapeziectomy but without the placement of the FlexHD acellular dermal matrix.

SUMMARY:
The objective of this study is to show that using FlexHD® (or HADM) to fill the empty space created by removal of the trapezium improves the subject's outcome and subsequent functionality of the basilar joint arthroplasty procedure.

DETAILED DESCRIPTION:
Subjects will be followed for 12 months post basilar joint arthroplasty procedure with an interposition arthroplasty technique using a spacer constructed from human acellular matrix (HADM). Their postoperative DASH scores, grip strength, pinch strength, pain scale scores, quality of life and trapezial space on radiographs are compared to their preoperative scores. Study visits will coincide with standard clinical course visits including: Pre-operative visits and follow-up visits at week 6, month 6, and year 1 post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female >18 years of age
* Be willing to undergo thumb basilar joint arthroplasty with the use of acellular dermal matrix
* Basilar Joint Arthritis Eaton Stage III or IV
* Be in good health other than the arthritis
* Have realistic expectations of surgical results
* Understand and be willing to follow all aspects of the study protocol and have signed and dated the IRB-approved Informed Consent Form and the Authorization for Use and Release of Health and Research Study Information (HIPAA) form prior to any study-related procedures being performed

Exclusion Criteria:

* Have collagen-vascular, connective tissue, or bleeding disorders
* Be a smoker or have smoked in last 2 months
* Have any disease, including uncontrolled diabetes, which is clinically known to impact wound healing ability
* Have regional sympathetic dystrophy
* Be pregnant, lactating or expecting to be within the next 24 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-08; Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Functionality | 12 months
  The objective of this study is to determine whether utilizing HADM will result in increased functionality measured by:
  * DASH score
  * Pinch and grip strength
  * Pain scale
  * Quality of life scores and
  * Trapezial space on radiographs at designated intervals during the post-operative period

CONTACTS AND LOCATIONS:
Overall Officials: David Kulber, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Department of Hand Surgery, Los Angeles, California, United States

REFERENCES:
- [Background] Ellis CV, Kulber DA. Acellular dermal matrices in hand reconstruction. Plast Reconstr Surg. 2012 Nov;130(5 Suppl 2):256S-269S. doi: 10.1097/PRS.0b013e318265a5cf. PMID 23096981
- [Background] Yao CA, Ellis CV, Cohen MJ, Kulber DA. Preserving the posttrapeziectomy space with a human acellular dermal matrix spacer: a pilot case series of patients with thumb carpometacarpal joint arthritis. Plast Reconstr Surg Glob Open. 2013 Nov 7;1(7):e65. doi: 10.1097/GOX.0b013e3182aa8793. eCollection 2013 Oct. PMID 25289260
- [Background] Gangopadhyay S, McKenna H, Burke FD, Davis TR. Five- to 18-year follow-up for treatment of trapeziometacarpal osteoarthritis: a prospective comparison of excision, tendon interposition, and ligament reconstruction and tendon interposition. J Hand Surg Am. 2012 Mar;37(3):411-7. doi: 10.1016/j.jhsa.2011.11.027. Epub 2012 Feb 3. PMID 22305824